CLINICAL TRIAL: NCT04635163
Title: Ideation Trajectories and Suicide Attempts in Adolescents With Psychiatric Disorders in the Maule Region. Chile
Brief Title: Ideation Trajectories and Suicide Attempts in Adolescents With Psychiatric Disorders in Chile
Status: Completed | Type: Observational
Sponsor: Universidad Católica del Maule (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Pablo Méndez-Bustos, Ph.D., Principal Investigator, Universidad Católica del Maule
Other Study IDs: University Catholic of Maule
Record Dates: First submitted 2020-10-22; First posted 2020-11-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Disorders; Suicide, Attempted
Keywords: Suicidal behavior; Psychiatric disorders; Adolescents
MeSH Terms: conditions — Mental Disorders; Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention — None intervention

SUMMARY:
This project seeks to evaluate the trajectories of suicidal ideation and attempts in adolescent patients with psychiatric disorders in secondary care controls in the Maule region, in relation to clinical factors (depressive symptoms, anxiety, stress, psychiatric comorbidity, mistreatment or abuse, history of psychiatric disorders and pharmacological treatments); psychological (parenting styles, impulsivity, barriers in seeking help and emotional regulation), and neuropsychological (executive function-decision making).

DETAILED DESCRIPTION:
Background

Adolescent suicide is a major problem in public health worldwide and due to the multi-dimensionality of factors involved (biological, genetic, psychiatric, economic, socio-demographic, family-related and cultural), its study is complex. Within the general population, the global suicide rate is 10.6 deaths for every 100,000 inhabitants (13.5 men and 7.7 women) and in the Americas it comes up to 9.8 deaths for every 100,000 inhabitants (15.1 men and 4.6 women). In Chile, the suicide rate is 10.6 deaths for every 100,000 inhabitants (17.2 men and 4.0 women) being above average regarding other countries in the Americas.

For adolescents, suicide is the second cause of premature death among people ranging from 15 to 29 and the third for the 15-19 age group. Also, within the group of 10 to 24 there are more deaths from suicide than traffic accidents, cancer, and cardiac diseases. In Chile, 60% of deaths among adolescents are caused by external reasons (suicide and homicide). Deaths to suicide among Chilean adolescents have presented a sustained increase in the last 15 years (55% between 1999-2005), being the second country within the Organization for Economic Co-operation and Development (OECD) with the highest percentage variation. In a recent study which compared the suicide rate among adolescents from 10 to 19 in countries belonging to the OECD, Chile had the fourth highest suicide rate with 5.36 deaths for every 100,000 inhabitants. When divided into sub-groups, Chile had the highest rates from 10 to 14 in both men and women with 2.23 deaths for every 100,000 inhabitants; and in the group of 15 to 19 the third highest rates in males and the fourth in females with 15.87 and 6.32 deaths for every 100,000 inhabitants, respectively.

Adolescence is a critical period of vulnerability for the development of suicidal behavior. During this stage, suicidal behavior shows unstable and fluctuating patterns; ideation without suicide attempts may appear, subjects can go from ideas to plans and make an attempt, there are those who try just once while others try repeatedly, and there are others who, in spite of their vulnerability, do not develop such behavior. Suicide rates vary according to gender and age, being higher among men than women, while ideation and suicide attempts are more frequent among women rather than men. It is estimated that for each completed suicide in young people, there are from 100 to 200 suicide attempts. Also, suicidal thoughts have been associated to later attempts and their repetition. It is estimated that a third of adolescents with suicidal thoughts will try during the following year. Evidence shows that lifetime the suicidal ideation rate is 12.1% in adolescents from 13 to 18; on the other hand, 7.4% of young people from 10 to 24 have reported at least one suicide attempt within the last 12 months with a greater prevalence of attempts among women (9.3%) than men (5.1%). In Chile, 23.7% of adolescents ranging from 13 to 18 presented suicidal ideation and 9% tried in the last 12 months.

The Chilean Health Ministry [MINSAL in Spanish] projected a rate of 12 deaths for every 100,000 inhabitants for adolescents from 10 to 19 for the year 2020. According to the sanitary objectives for the 2011-2020 decade, the MINSAL got determined to diminish this projected rate by 15%. However, in Chile there are still various limitations and challenges regarding the study of suicidal behavior among adolescent population. Considering the risk of onset of suicidal thoughts and attempts during adolescence and the variability in their evolution, it becomes necessary to make an early and timely identification of high-risk clinical sub-groups. The analysis of both their patterns along a timeframe and the influence and interaction of specific factors could meet such objective.

The present study aims to evaluate the trajectories of suicidal ideation and attempts in adolescents with psychiatric disorders being treated within the public health system of the Maule Region, Chile, in relation to clinical, psychological, and neuropsychological factors.

Specific objectives

1. Identify patterns of change in the trajectories of suicidal ideation and attempts based on the type of psychiatric disorder.
2. Identify clinical, psychological, and neuropsychological factors for suicide ideation and attempts during the follow-up period.
3. To determine the predictive value of clinical, psychological, and neuropsychological factors on the course of suicidal ideation and attempts in adolescent psychiatric patients.
4. To evaluate the interaction of clinical, psychological, and neuropsychological factors and their influence on the course of suicidal ideation and attempts in adolescent psychiatric patients.
5. Identify and characterize groups of adolescent patients with psychiatric disorders, according to the course of ideation and suicide attempts.
6. Identify and characterize groups of adolescent patients with psychiatric disorders, according to repetition of suicide attempts.

Study design. A prospective naturalist study of repeated measurements with a single group.

Instruments

1. Columbia University Rating Scale on the Intensity of Suicidal Ideas (C-SSRS Chile / Spanish 5.1)
2. Barratt Impulsivity Scale
3. Emotional Regulation Difficulties Scale (DERS-E)
4. Depression, Anxiety and Stress abbreviated Scale (DASS-21)
5. Insomnia Severity Index (ISI)
6. Brief Parental Scale (BPS).
7. General Help Seeking Questionnaire for mental health problems in adolescents (GHSQ)
8. Iowa Gambling Task (IGT).

Procedure and Application

Dissemination of the study will be made along with mental health teams in hospitals, Community Centers for Mental Health (COSAM) and Family Health Centers (CESFAM) of the Maule Region. After the study has initiated, a registry will be made of the patients who attend the Mental Health units during the first 6 months. Patients shall be contacted by a member of the research team and invited to participate, informing them in written and verbally about the essential aspects of the research, its objective, benefits, and clinical implications. Afterwards, their informed consent shall be requested, which must be signed by the mother, father, or responsible tutor for participants under 18. Selected patients shall be assessed using the protocol made up by the instruments before mentioned at three moments during the study: an initial evaluation, then at 6-8 months, and the final evaluation one year after the second measurement. Medical records will be analyzed to obtain data regarding medical history (psychiatric and medical diagnose, hospitalization, treatments, among others) and a socio-demographic questionnaire is to be applied. Also, family-related background is to be obtained regarding records of mental disease and suicidal behavior.

During the research and the follow-up period (24 months), the responsible researcher shall arrange clinical meetings with the team or professionals (medics or psychologists) of the adolescents under study.

Statistical analysis and expected results

Initially, different exploratory analysis will be carried out with the goal of obtaining a first approximation to the data and spot out possible coding errors. Then, analysis shall be made regarding reliability and validity for each of the instruments constituting the protocol. Modeling techniques will also be implemented with the objective of analyzing the information gathered from an explicative and predictive perspective, exploring the adjustment levels of data in the models being tested.

Finally, from the latent class analyzes, we will seek to identify change trajectories in relation to the variables studied, based on the following hypotheses:

1. High levels of suicidal ideation at first measurement, predicts a higher likelihood of suicide attempts during the follow-up period.
2. Adolescents with suicidal ideation and previous attempts will be more likely to repeat than those with a single attempt.
3. Adolescents with less emotional regulation, poor parental styles, high levels of impulsivity and a history of self-harm have an irregular course of suicidal thoughts and ask for less help in dealing with their problems.
4. Adolescents with a history of previous suicide attempts, psychiatric comorbidity, and impaired decision-making ability, have a greater severity of suicidal ideas and more likely to repeat a suicide attempt than those without these characteristics.

Ethical review

The research project was approved by the Ethics Committee of the Maule Health Service and by the Scientific Ethics Committee of the Universidad Católica del Maule de Chile, meeting principles established by the Universal Declaration of Human Rights, international regulations of the Council for International Organizations of Medical Sciences (CIOMS) and Law 20.120 regarding scientific research involving human beings in Chile. Also, the authors declare that necessary ethical safeguards have been adopted for working with people, as proposed in the Helsinki declaration and the Belmont report.

Discussion

Adolescent suicide is the consequence of a complex interaction among genetic, biological, psychiatric, psychological, social, and cultural factors. Though there is consensus regarding the importance of elaborating more effective interventions for reducing suicide risk among adolescents, there still are many limitations and challenges in the detection and early and timely prevention of suicidal thoughts and attempts.

A review of the existing evidence have pointed out that models proposed in the last 50 years present a low predictive capacity and that risk factor categories have become homogeneous, being incapable of identifying specific groups of variables associated to the different types of suicidal behavior.

On the other hand, it is paradoxical that about 82% of scientific production comes from North America and Europe, considering that countries such as China and India account for almost half of suicides worldwide, and given the sustained increase in suicide rates in Latin America, where several countries exceed the European average. It is necessary to promote more studies in these territories and identify cultural and local variables that can improve the understanding of this public health problem.

Considering the risk of onset of ideation and suicidal attempts during adolescence and the variability in their evolution, it becomes necessary to early and timely identify vulnerable groups by means of different methodological approaches. This way, their study requires methodological approaches that allow overcoming detected weaknesses, through specific explicative models which enable a more in-depth comprehension of their development.

The methodology proposed for this study will seek to overcome the limitations of cross-sectional and retrospective studies by identifying patterns of suicidal thoughts and behaviors for a specified period and of the influence and interactions of specific variables.

On the other hand, though the number of total questions of the protocol may seem high, the selected questionnaires present a form of short answers which are easy to comprehend. Also, each questionnaire will be applied by a trained research assistant (psychologist) and each question shall be read to the adolescent to ensure understanding and quality of the answer.

Although the use of protocols in clinical practice has been questioned due to their low predictive capacity, their use can improve efficiency and consistency in decision making, allowing the elaboration of an individualized treatment plan and a better risk management.

Finally, deaths by self-inflicted injuries are irregularly distributed around the world, 79% of suicides occur in low and mid income countries but, in spite of the importance of considering these regional variations and the differentiation of risk factors according to the context, most researches take place in high income countries (Europe and North America) where the risk of suicide is lower.

This study also seeks to overcome this weakness so as to allow comparing and identifying differentiating aspects of suicidal behavior in adolescents, which will contribute to improve the understanding of this problem and to elaborate interventions focused on sub-clinical groups with higher risk, also considering cultural and local variables.

ELIGIBILITY:
Inclusion criteria:

* Adolescents between 15 and 19 years old
* Diagnosed with psychiatric disorder
* With and without suicidal ideation
* With and without suicide attempts
* With the ability to read and write
* Those who give their assent, in addition to an informed consent signed by their mother and / or father or legal representative

Exclusion criteria

* Adolescents who do not have the ability to read and / or write.
* Those who refuse to participate in the study, whose mother and / or father or legal representative do not give their consent
* Suffering from a disabling medical illness and / or active psychotic symptoms

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents of both genders will be selected utilizing a non-probability purposive sampling, ranging from 15 to 19 years of age and diagnosed with a psychiatric disorder with or without ideation and suicidal attempts, being under treatment in Mental Health units in hospitals and Health Centers in the Maule Region, with capacity for reading and writing, and not presenting an disabling medical illness and/or active psychotic symptomatology.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
High levels of suicidal ideation and likelihood of suicide attempts during the follow-up period | 3 years
  High levels of suicidal ideation at first measurement, predicts a higher likelihood of suicide attempts during the follow-up period.
Suicidal ideation and previous attempts versus single attempt | 3 years
  Adolescents with suicidal ideation and previous attempts will be more likely to repeat than those with a single attempt.
Clinical and psychological factors, predispose irregular course of suicidal thoughts and scant seek for help. | 3 years
  Adolescents with less emotional regulation, poor parenting styles, high levels of impulsivity and a history of self-harm will have significant differences in levels of suicidal ideation during the follow-up period (3 measurements) and more than 60% of them will report that they do not seek help to deal with your mental health problems.
Severity of suicidal ideation according to psychiatric comorbidity, impaired decision-making capacity, and previous suicide attempts. | 3 years
  Adolescents with previous suicide attempts, psychiatric comorbidity, and impaired decision-making capacity, have a greater severity of suicidal ideas, and consequently, are more likely to repeat a suicide attempt than those without these characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- University Catholic Maule. Chile, Talca, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasserman D, Rihmer Z, Rujescu D, Sarchiapone M, Sokolowski M, Titelman D, Zalsman G, Zemishlany Z, Carli V; European Psychiatric Association. The European Psychiatric Association (EPA) guidance on suicide treatment and prevention. Eur Psychiatry. 2012 Feb;27(2):129-41. doi: 10.1016/j.eurpsy.2011.06.003. Epub 2011 Dec 1. PMID 22137775
- [Background] Miranda R, Shaffer D. Understanding the suicidal moment in adolescence. Ann N Y Acad Sci. 2013 Nov;1304:14-21. doi: 10.1111/nyas.12291. Epub 2013 Oct 18. PMID 24138124
- [Background] Schrijvers DL, Bollen J, Sabbe BG. The gender paradox in suicidal behavior and its impact on the suicidal process. J Affect Disord. 2012 Apr;138(1-2):19-26. doi: 10.1016/j.jad.2011.03.050. Epub 2011 May 6. PMID 21529962
- [Result] Bachmann S. Epidemiology of Suicide and the Psychiatric Perspective. Int J Environ Res Public Health. 2018 Jul 6;15(7):1425. doi: 10.3390/ijerph15071425. PMID 29986446
- [Result] Shain B; COMMITTEE ON ADOLESCENCE. Suicide and Suicide Attempts in Adolescents. Pediatrics. 2016 Jul;138(1):e20161420. doi: 10.1542/peds.2016-1420. PMID 27354459
- [Result] Roh BR, Jung EH, Hong HJ. A Comparative Study of Suicide Rates among 10-19-Year-Olds in 29 OECD Countries. Psychiatry Investig. 2018 Apr;15(4):376-383. doi: 10.30773/pi.2017.08.02. Epub 2018 Feb 28. PMID 29486551
- [Result] Breton JJ, Tousignant M, Bergeron L, Berthiaume C. Informant-specific correlates of suicidal behavior in a community survey of 12- to 14-year-olds. J Am Acad Child Adolesc Psychiatry. 2002 Jun;41(6):723-30. doi: 10.1097/00004583-200206000-00012. PMID 12049447
- [Result] Nock MK, Green JG, Hwang I, McLaughlin KA, Sampson NA, Zaslavsky AM, Kessler RC. Prevalence, correlates, and treatment of lifetime suicidal behavior among adolescents: results from the National Comorbidity Survey Replication Adolescent Supplement. JAMA Psychiatry. 2013 Mar;70(3):300-10. doi: 10.1001/2013.jamapsychiatry.55. PMID 23303463
- [Result] McLoughlin AB, Gould MS, Malone KM. Global trends in teenage suicide: 2003-2014. QJM. 2015 Oct;108(10):765-80. doi: 10.1093/qjmed/hcv026. Epub 2015 Jan 31. PMID 25638789
- [Result] Miranda R, De Jaegere E, Restifo K, Shaffer D. Longitudinal follow-up study of adolescents who report a suicide attempt: aspects of suicidal behavior that increase risk of a future attempt. Depress Anxiety. 2014 Jan;31(1):19-26. doi: 10.1002/da.22194. Epub 2013 Sep 18. PMID 24105789
- [Result] Annor FB, Clayton HB, Gilbert LK, Ivey-Stephenson AZ, Irving SM, David-Ferdon C, Kann LK. Sexual Orientation Discordance and Nonfatal Suicidal Behaviors in U.S. High School Students. Am J Prev Med. 2018 Apr;54(4):530-538. doi: 10.1016/j.amepre.2018.01.013. Epub 2018 Feb 21. PMID 29449136
- [Derived] Mendez-Bustos P, Fuster-Villaseca J, Lopez-Castroman J, Jimenez-Solomon O, Olivari C, Baca-Garcia E. Longitudinal trajectories of suicidal ideation and attempts in adolescents with psychiatric disorders in Chile: study protocol. BMJ Open. 2022 Feb 22;12(2):e051749. doi: 10.1136/bmjopen-2021-051749. PMID 35193905
- See also: Suicidal behavior in children and adolescents: Epidemiology and risk factors — https://www.uptodate.com/contents/suicidal-behavior-in-children-and-adolescents-epidemiology-and-risk-factors?topicRef=4867
- See also: Suicide, Keys facts — https://www.who.int/news-room/fact-sheets/detail/suicide
- See also: Programa nacional de prevención del suicidio: orientaciones para su implementación — https://www.minsal.cl/sites/default/files/Programa_Nacional_Prevencion.pdf
- See also: Epidemiology of Suicidal and Risk-Taking Behavior — https://www.cambridge.org/core/journals/european-psychiatry/article/s3901-epidemiology-of-suicidal-and-risktaking-behavior/EBA2D1F739AC40E6416BB20036090168
- See also: Intento de suicidio y factores de riesgo en una muestra de adolescentes escolarizados de Chile — http://revistas.uned.es/index.php/RPPC/article/view/16170
- See also: Estrategia Nacional de Salud para el cumplimiento de los objetivos sanitarios de la década 2011-2020 — https://www.minsal.cl/portal/url/item/c4034eddbc96ca6de0400101640159b8.pdf